CLINICAL TRIAL: NCT02835716
Title: Pre-Clinical Alzheimer's (ALZ) Diagnosis (PCD) = Optimum Outcomes (OO)
Brief Title: Pre-Clinical (Alzheimers) Diagnosis PCD = Optimum Outcomes OO
Acronym: PCD=OOALZ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Millennium Magnetic Technologies, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: PCD=OO ALZ
Record Dates: First submitted 2016-07-10; First posted 2016-07-18 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Alzheimer Disease
Keywords: Phosphodiesterase type 4 inhibitor; ustekinumab; secukinumab; P40 subunit; Interleukin IL-12; Interleukin IL-23; Apoprotein e4; Interleukin IL-17A
MeSH Terms: conditions — Alzheimer Disease | interventions — Roflumilast; Ustekinumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: roflumilast — DALIRESP is used in adults with severe chronic obstructive pulmonary disease (COPD) to decrease the number of flare-ups or the worsening of COPD symptoms (exacerbations
  Other Names: Daliresp
Biological: ustekinumab — STELARA is approved to treat adults 18 years and older with moderate or severe plaque psoriasis that involves large areas or many areas of their body
  Other Names: Stelara

SUMMARY:
This Observational protocol will attempt to verify two recent and very critical concepts in ALZ Clinical Research by studying high-risk individuals who already are taking medications which may prevent the onset of ALZ.

* It may be possible to determine the future development of ALZ in a preclinical state in a cognitively normal but high risk individual at least 18-24 months before any symptoms develop of cognitive impairment.
* Early treatment of these cognitively normal high-risk persons with subclinical pre-ALZ can prevent of delay the occurrence and severity of ALZ.

Caveats

Neither this protocol nor the fMRI imaging are designed or intended to diagnose or treat ALZ, nor develop or use medications or diagnostic neuroimaging outside of already approved and accepted parameters. Persons who volunteer to be study subjects in this observational protocol will be under the care of their primary care / specialty physician, who will order tests and treatments as they see appropriate.

Although there is a very large body of peer-reviewed scientific literature demonstrating that certain functional MRI patterns are associated with certain neurologic conditions, the utilization of fMRI for the evaluation of neurologic disorders is still considered an emerging science and therefore in the investigational stage. Although this protocol will report on brain patterns of certain neurologic conditions such as cognitive impairment and Alzheimer's disease, based on patterns published in peer-reviewed journals, such findings are not considered stand alone or diagnostic per se and should always be considered by the PMD in conjunction with the patient's clinical condition. These data should only be used as additional information to add to the PMD's diagnostic impression.

DETAILED DESCRIPTION:
Prospective observational study participants age 50-75 years are identified who are currently (<1 month) taking or will soon (within 3 months) start taking study medications of interest thru their own physician.

Prospective observational study participants are explained how persons can be cognitively normal but at high risk for developing clinical ALZ, and that this risk can be prospectively identified.

They are advised that there is some rationale that medications they are or will soon be taking may have a protective effect in delaying the onset of ALZ, and that protective effect can be monitored.

They are asked if they would like to participate in a protocol that monitors their prospective risk for developing ALZ short term, and whether certain of their prescribed medications may have a protective effect. Those who are accepting to be participants are then enrolled in the study.

Enrollees are tested for risk factors for having pre-clinical ALZ. Individuals identified as being at risk at baseline are followed at 6 month intervals for a 24 month period using psychometric testing and functional neuroimaging. Their maintenance of cognitive stability or cognitive decline is monitored while under the care of their PMD and while taking medications of interest.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 75 years old,
* Normal baseline cognitive function by standard psychometric testing.
* Able to privately fund psychometric and neuroimaging studies if not covered by their insurance,
* Able to give written Informed Consent,
* Ascent for collaboration by their primary care or specialty physician,
* Currently taking (<1 month) or planning to take (within the next 3 months) medications which are identified in the study group of interest, prescribed by and under the care of a PMD or specialty physician.

Exclusion Criteria:

• Inability to undergo MR Imaging : Claustrophobia, certain metal implants,

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults at high risk of developing ALZ within 18-48 months but are currently cognitively normal for their age sex matching group. Risk factors include parents with a history of ALZ, and/or positive APOE4 alleles.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Develop Cognitive Decline | 18-24 month
  Cognitive decline is defined as a reduction from baseline performance within each individual of at least one standard deviation (SD) on at least one of the three principal outcome indices (DRS-2, RAVLT Sum of Trials 1-5 [T1- 5], RAVLT Delayed Recall [DR]).

CONTACTS AND LOCATIONS:
Overall Officials: Donald H Marks, MD PhD, Principal Investigator — MMT
Locations (1):
- Millennium Magnetic Technologies, LLC, Westport, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bangen KJ, Restom K, Liu TT, Wierenga CE, Jak AJ, Salmon DP, Bondi MW. Assessment of Alzheimer's disease risk with functional magnetic resonance imaging: an arterial spin labeling study. J Alzheimers Dis. 2012;31 Suppl 3(0):S59-74. doi: 10.3233/JAD-2012-120292. PMID 22531427
- [Background] Caltagirone C, Ferrannini L, Marchionni N, Nappi G, Scapagnini G, Trabucchi M. The potential protective effect of tramiprosate (homotaurine) against Alzheimer's disease: a review. Aging Clin Exp Res. 2012 Dec;24(6):580-7. doi: 10.3275/8585. Epub 2012 Sep 5. PMID 22961121
- [Background] Cavedo E, Lista S, Khachaturian Z, Aisen P, Amouyel P, Herholz K, Jack CR Jr, Sperling R, Cummings J, Blennow K, O'Bryant S, Frisoni GB, Khachaturian A, Kivipelto M, Klunk W, Broich K, Andrieu S, de Schotten MT, Mangin JF, Lammertsma AA, Johnson K, Teipel S, Drzezga A, Bokde A, Colliot O, Bakardjian H, Zetterberg H, Dubois B, Vellas B, Schneider LS, Hampel H. The Road Ahead to Cure Alzheimer's Disease: Development of Biological Markers and Neuroimaging Methods for Prevention Trials Across all Stages and Target Populations. J Prev Alzheimers Dis. 2014 Dec;1(3):181-202. doi: 10.14283/jpad.2014.32. PMID 26478889
- [Background] Chincarini A, Bosco P, Calvini P, Gemme G, Esposito M, Olivieri C, Rei L, Squarcia S, Rodriguez G, Bellotti R, Cerello P, De Mitri I, Retico A, Nobili F; Alzheimer's Disease Neuroimaging Initiative. Local MRI analysis approach in the diagnosis of early and prodromal Alzheimer's disease. Neuroimage. 2011 Sep 15;58(2):469-80. doi: 10.1016/j.neuroimage.2011.05.083. Epub 2011 Jun 16. PMID 21718788
- [Background] Chiang K, Koo EH. Emerging therapeutics for Alzheimer's disease. Annu Rev Pharmacol Toxicol. 2014;54:381-405. doi: 10.1146/annurev-pharmtox-011613-135932. PMID 24392696
- [Background] Chao S, Roberts JS, Marteau TM, Silliman R, Cupples LA, Green RC. Health behavior changes after genetic risk assessment for Alzheimer disease: The REVEAL Study. Alzheimer Dis Assoc Disord. 2008 Jan-Mar;22(1):94-7. doi: 10.1097/WAD.0b013e31815a9dcc. PMID 18317253
- [Background] Deardorff WJ, Grossberg GT. Targeting neuroinflammation in Alzheimer's disease: evidence for NSAIDs and novel therapeutics. Expert Rev Neurother. 2017 Jan;17(1):17-32. doi: 10.1080/14737175.2016.1200972. Epub 2016 Jun 24. PMID 27293026
- [Background] Garcia-Osta A, Cuadrado-Tejedor M, Garcia-Barroso C, Oyarzabal J, Franco R. Phosphodiesterases as therapeutic targets for Alzheimer's disease. ACS Chem Neurosci. 2012 Nov 21;3(11):832-44. doi: 10.1021/cn3000907. Epub 2012 Oct 1. PMID 23173065
- [Background] Galluzzi S, Marizzoni M, Babiloni C, Albani D, Antelmi L, Bagnoli C, Bartres-Faz D, Cordone S, Didic M, Farotti L, Fiedler U, Forloni G, Girtler N, Hensch T, Jovicich J, Leeuwis A, Marra C, Molinuevo JL, Nobili F, Pariente J, Parnetti L, Payoux P, Del Percio C, Ranjeva JP, Rolandi E, Rossini PM, Schonknecht P, Soricelli A, Tsolaki M, Visser PJ, Wiltfang J, Richardson JC, Bordet R, Blin O, Frisoni GB; PharmaCog Consortium. Clinical and biomarker profiling of prodromal Alzheimer's disease in workpackage 5 of the Innovative Medicines Initiative PharmaCog project: a 'European ADNI study'. J Intern Med. 2016 Jun;279(6):576-91. doi: 10.1111/joim.12482. Epub 2016 Mar 4. PMID 26940242
- [Background] Griffin WS. Neuroinflammatory cytokine signaling and Alzheimer's disease. N Engl J Med. 2013 Feb 21;368(8):770-1. doi: 10.1056/NEJMcibr1214546. No abstract available. PMID 23425171
- [Background] Gurney ME, D'Amato EC, Burgin AB. Phosphodiesterase-4 (PDE4) molecular pharmacology and Alzheimer's disease. Neurotherapeutics. 2015 Jan;12(1):49-56. doi: 10.1007/s13311-014-0309-7. PMID 25371167
- [Background] Christensen KD, Roberts JS, Whitehouse PJ, Royal CD, Obisesan TO, Cupples LA, Vernarelli JA, Bhatt DL, Linnenbringer E, Butson MB, Fasaye GA, Uhlmann WR, Hiraki S, Wang N, Cook-Deegan R, Green RC; REVEAL Study Group*. Disclosing Pleiotropic Effects During Genetic Risk Assessment for Alzheimer Disease: A Randomized Trial. Ann Intern Med. 2016 Feb 2;164(3):155-63. doi: 10.7326/M15-0187. Epub 2016 Jan 26. PMID 26810768
- [Background] Green RC, Christensen KD, Cupples LA, Relkin NR, Whitehouse PJ, Royal CD, Obisesan TO, Cook-Deegan R, Linnenbringer E, Butson MB, Fasaye GA, Levinson E, Roberts JS; REVEAL Study Group. A randomized noninferiority trial of condensed protocols for genetic risk disclosure of Alzheimer's disease. Alzheimers Dement. 2015 Oct;11(10):1222-30. doi: 10.1016/j.jalz.2014.10.014. Epub 2014 Dec 9. PMID 25499536
- [Background] Haller S, Nguyen D, Rodriguez C, Emch J, Gold G, Bartsch A, Lovblad KO, Giannakopoulos P. Individual prediction of cognitive decline in mild cognitive impairment using support vector machine-based analysis of diffusion tensor imaging data. J Alzheimers Dis. 2010;22(1):315-27. doi: 10.3233/JAD-2010-100840. PMID 20847435
- [Background] Heckman PR, Wouters C, Prickaerts J. Phosphodiesterase inhibitors as a target for cognition enhancement in aging and Alzheimer's disease: a translational overview. Curr Pharm Des. 2015;21(3):317-31. doi: 10.2174/1381612820666140826114601. PMID 25159073
- [Background] Li NC, Lee A, Whitmer RA, Kivipelto M, Lawler E, Kazis LE, Wolozin B. Use of angiotensin receptor blockers and risk of dementia in a predominantly male population: prospective cohort analysis. BMJ. 2010 Jan 12;340:b5465. doi: 10.1136/bmj.b5465. PMID 20068258
- [Background] Langbaum JB, Fleisher AS, Chen K, Ayutyanont N, Lopera F, Quiroz YT, Caselli RJ, Tariot PN, Reiman EM. Ushering in the study and treatment of preclinical Alzheimer disease. Nat Rev Neurol. 2013 Jul;9(7):371-81. doi: 10.1038/nrneurol.2013.107. Epub 2013 Jun 11. PMID 23752908
- [Background] Lazarczyk MJ, Hof PR, Bouras C, Giannakopoulos P. Preclinical Alzheimer disease: identification of cases at risk among cognitively intact older individuals. BMC Med. 2012 Oct 25;10:127. doi: 10.1186/1741-7015-10-127. PMID 23098093
- [Background] Peters KR, Lynn Beattie B, Feldman HH, Illes J. A conceptual framework and ethics analysis for prevention trials of Alzheimer Disease. Prog Neurobiol. 2013 Nov;110:114-23. doi: 10.1016/j.pneurobio.2012.12.001. Epub 2013 Jan 21. PMID 23348495
- [Background] Riedel WJ. Preventing cognitive decline in preclinical Alzheimer's disease. Curr Opin Pharmacol. 2014 Feb;14:18-22. doi: 10.1016/j.coph.2013.10.002. Epub 2013 Nov 13. PMID 24565007
- [Background] Rizk-Jackson A, Insel P, Petersen R, Aisen P, Jack C, Weiner M. Early indications of future cognitive decline: stable versus declining controls. PLoS One. 2013 Sep 9;8(9):e74062. doi: 10.1371/journal.pone.0074062. eCollection 2013. PMID 24040166
- [Background] Zhou Y, Tan C, Wen D, Sun H, Han W, Xu Y. The Biomarkers for Identifying Preclinical Alzheimer's Disease via Structural and Functional Magnetic Resonance Imaging. Front Aging Neurosci. 2016 Apr 27;8:92. doi: 10.3389/fnagi.2016.00092. eCollection 2016. No abstract available. PMID 27199739
- [Background] Vernarelli JA, Roberts JS, Hiraki S, Chen CA, Cupples LA, Green RC. Effect of Alzheimer disease genetic risk disclosure on dietary supplement use. Am J Clin Nutr. 2010 May;91(5):1402-7. doi: 10.3945/ajcn.2009.28981. Epub 2010 Mar 10. PMID 20219963
- [Background] Vom Berg J, Prokop S, Miller KR, Obst J, Kalin RE, Lopategui-Cabezas I, Wegner A, Mair F, Schipke CG, Peters O, Winter Y, Becher B, Heppner FL. Inhibition of IL-12/IL-23 signaling reduces Alzheimer's disease-like pathology and cognitive decline. Nat Med. 2012 Dec;18(12):1812-9. doi: 10.1038/nm.2965. Epub 2012 Nov 25. PMID 23178247
- [Background] Woodard JL, Seidenberg M, Nielson KA, Smith JC, Antuono P, Durgerian S, Guidotti L, Zhang Q, Butts A, Hantke N, Lancaster M, Rao SM. Prediction of cognitive decline in healthy older adults using fMRI. J Alzheimers Dis. 2010;21(3):871-85. doi: 10.3233/JAD-2010-091693. PMID 20634590
- [Background] Xekardaki A, Rodriguez C, Montandon ML, Toma S, Tombeur E, Herrmann FR, Zekry D, Lovblad KO, Barkhof F, Giannakopoulos P, Haller S. Arterial spin labeling may contribute to the prediction of cognitive deterioration in healthy elderly individuals. Radiology. 2015 Feb;274(2):490-9. doi: 10.1148/radiol.14140680. Epub 2014 Oct 7. PMID 25291458
- See also: Ustekinumab New Drug Therapy for Cognitive Decline resulting from Neuroinflammatory Cytokine Signaling and Alzheimer's Disease — https://pharmaceuticalintelligence.com/2013/02/27/ustekinumab-new-drug-therapy-for-cognitive-decline-resulting-from-neuroinflammatory-cytokine-signaling-and-alzheimers-disease/